CLINICAL TRIAL: NCT02093195
Title: Phase Ⅱ Study of Bosentan in the Treatment of Stable Severe Chronic Obstructive Pulmonary Disease Patients
Brief Title: Study of Bosentan in the Treatment of Stable Severe Chronic Obstructive Pulmonary Disease Patients
Acronym: BTCOPD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Shengqing Li, Associate Chief Physician, Associate Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTCOPD-2014226
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Treatment, COPD, bosentan
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Bosentan; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bosentan (Experimental): Bosentan,125mg,po,bid combined with inhaled Symbicort turbuhaler, 320/9μg, bid.
  Interventions: Drug: Bosentan; Drug: Symbicort turbuhaler
- Control (Active Comparator): Inhaled Symbicort turbuhaler, 320/9μg, bid.
  Interventions: Drug: Symbicort turbuhaler

INTERVENTIONS:
Drug: Bosentan
  Arms: Bosentan
Drug: Symbicort turbuhaler

SUMMARY:
Present treatment for chronic obstructive pulmonary disease (COPD) has a certain role in reducing COPD exacerbation and hospitalization, improving the life quality, and postponing the lung function decline. But for some patients with severe COPD, current treatment only partially alleviates the symptoms and has little role in the lung function decline. In this randomized, multicenter study, the investigators evaluate the safety and efficacy of bosentan in the treatment of grade Ⅲ or Ⅳ COPD patients with pulmonary hypertension detected by echocardiography. The primary endpoint is the frequency of COPD exacerbation, and the secondary endpoint includes changes of lung function, 6-min-walk distance (6-MWD), SGRQ score and mMRC/CAT score.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75
* Gold Ⅲ or Ⅳ stable COPD
* Pulmonary hypertension detected by echocardiography

Exclusion Criteria:

* Acute exacerbation of chronic obstructive pulmonary disease
* Untreated obstructive sleep apnea
* Restrictive (total lung capacity<60% predicted) lung disease
* Portal hypertension
* Chronic liver disease
* Transaminase increased to normal line more than 3 times; total bilirubin increased 2 times more than the upper limit of the normal value
* Left-sided or unrepaired congenital heart disease
* Patients with other serious heart diseases
* Patients with 1, 2, 4 and 5 categories of pulmonary hypertension
* Unable to complete the 6 minutes walk test
* Patients receiving other endothelin receptor antagonists
* No cooperation to complete

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of COPD Exacerbation | 12 months

SECONDARY OUTCOMES:
6-min-walk distance (6-MWD) | 12 months
Lung Function | 12 months
mMRC/CAT score | 12 months
SGRQ score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shengqing Li, MD, PhD, Principal Investigator — The department of pulmonary and critical care medicine, Xijing hospital
Locations (5):
- China (5):
  - The second affiliated hospital of xi'an jiaotong university, Xi'an, Shaanxi
  - The department of pulmonary and critical care medicine, Xijing hospital, Xi'an, Shaanxi
  - The department of pulmonary and critical care medicine, Tangdou hospital, Xi'an, Shaanxi
  - The first affiliated hospital of xi'an jiaotong university, Xi'an, Shaanxi
  - Shaanxi Provincial People'S Hospital, Xi'an, Shaanxi